CLINICAL TRIAL: NCT02920541
Title: Phase I Dose-escalation Study of the Orally Administered Selective Bcl-2 Inhibitor S 055746 as Monotherapy for the Treatment of Patients With Acute Myeloid Leukaemia (AML) or High or Very High Risk Myelodysplastic Syndrome (MDS)
Brief Title: Dose-escalation Study of Oral Administration of S 055746 in Patients With Acute Myeloid Leukaemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL1-055746-002; 2014-002559-24 (EudraCT Number); ISRCTN73586707 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2016-08-23; First posted 2016-09-30 (Estimated); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Acute Myeloid Leukaemia (AML); Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- S 055746 (Experimental)
  Interventions: Drug: S 055746

INTERVENTIONS:
Drug: S 055746 — S 055746, per os administration, from 50 to 2000 mg once a day during a 21-day cycle. Participants will receive 21-day cycles of treatment until a discontinuation criterion is met.

SUMMARY:
The purpose of this study is to determine the safety profile and tolerability of S 055746 in patients with AML, and high or very high risk MDS, in terms of Dose-Limiting Toxicities (DLTs), Maximum Tolerated Dose (MTD) and determine the Recommended Phase 2 Dose (RP2D) through safety profile (DLT, MTD), PK profile, PD profile and preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Women or men aged >= 18 years
* Patients with cytologically confirmed and documented de novo, secondary or therapy-related AML excluding acute promyelocytic leukaemia:

  * with relapsed or refractory disease or
  * > or = 65 years not previously treated for AML, who are not candidates for intensive chemotherapy or not candidates for standard chemotherapy
* Patients with cytologically confirmed and documented MDS or non proliferative Chronic Myelomonocytic Leukaemia (CMML) in relapse or refractory after previous treatment line including at least one hypomethylating agent therapy:

  * with high or very high risk MDS and without established alternative therapy
  * transformed to AML and without established alternative therapy
* Ability to swallow oral tablet(s)
* World Health Organization (WHO) performance status 0-2
* Circulating white blood cells < or = 30 x 10^9 /L and < or = 13 x10^9 for non proliferative CMML
* Adequate renal and hepatic functions
* Negative serum pregnancy test within 7 days prior to the first day of study drug administration
* Patients must use effective contraception
* Written informed consent

Exclusion Criteria:

* Foreseeable poor compliance to the study procedures
* Legally incapacitated person under guardianship or trusteeship
* Pregnant or breast-feeding women
* Participation in therapeutic interventional study involving investigational drug intake at the same time or within 2 weeks or at least 5 half-lives or patient already enrolled
* Previous treatment with a BH3 mimetic
* Patients who have not recovered to baseline or CTCAE< or = Grade 1 from toxicity due to all prior therapies received for the studied disease
* Any previous anti-leukaemic treatment for the studied disease within at least 5 half-lives or 2 weeks (hydroxycarbamide permitted)
* Any radiotherapy within 4 weeks before first intake (except palliative radiotherapy at localized lesions)
* Major surgery within 3 weeks before first intake of S 055746
* Allogenic stem cell transplant within 6 months before the first intake of S 055746 and for patients who still need immunosuppressive treatment
* Leukaemic leptomeningeal or leukaemic central nervous system involvement
* Concomitant uncontrolled infection, organ dysfunction or medical disease likely to interfere with evaluation of S 055746 safety or study outcome
* Human immunodeficiency virus (HIV) infection, hepatitis B or active hepatitis C infection
* Within 6 months prior to the first intake of S 055746, history of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, and/or stenting, ischemic/haemorrhagic stroke, atrial fibrillation, digestive haemorrhagic risk, deep venous/arterial thromboembolic complication or bleeding diathesis
* Decreased Left Ventricular Ejection Fraction (LVEF)
* QTcF prolongation
* Patients who are receiving QT prolonging drug
* Coagulopathies with increased risk of bleeding complications
* Other malignancy within 2 years prior to the first intake
* Strong or moderate CYP3A4 inhibitors or inducers (treatment, food or drink products) within 7 days prior to the first intake
* Treatment highly metabolised by the CYP3A4 or CYP2D6 and/or with a narrow therapeutic index, multi-enzymes and/or OATP and/or P-gp substrates or herbal products within 7 days prior to the first intake.
* Patients receiving proton pump inhibitor
* Patients having received anticoagulant oral drugs, aspirin > 325 mg/day and antiplatelets within 7 days prior to first S 055746 intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-01; Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | During cycle 1 (21 days)
  MTD is the highest drug dosage that is unlikely (<25% posterior probability) to cause DLT in more than 33% of the treated patients in the first cycle of S 055746 treatment.
Incidence of Adverse Events (AEs) | From first dose until 30 days after the last dose intake
  Characterized by severity and seriousness of AEs, laboratory abnormalities and other safety parameters such as electrocardiogram (ECG) changes

SECONDARY OUTCOMES:
Plasma concentration of S 055746 | Pre-dose on Cycle 1 Day 1 (C1D1), C1D2, C1D3, C1D8, C1D9, C2D1 ; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10-12 hours post-dose on C1D1, C1D8
The pharmacokinetic (PK) profile of S 055746: Area Under the Curve [AUC] | Pre-dose on Cycle 1 Day 1 (C1D1), C1D2, C1D3, C1D8, C1D9, C2D1 ; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10-12 hours post-dose on C1D1, C1D8
The PK profile of S 055746: Maximal Concentration [Cmax] | Pre-dose on Cycle 1 Day 1 (C1D1), C1D2, C1D3, C1D8, C1D9, C2D1 ; 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10-12 hours post-dose on C1D1, C1D8
Best Response Rate (BRR) | Up to study completion (maximum of 3 years)
Progression Free Survival (PFS) | From date of inclusion until the date of progression or date of death, whichever occurs first, assessed up to study completion (maximum of 3 years)
Event Free Survival (EFS) | From date of inclusion until the date of progression or date of death or discontinuation of treatment, whichever occurs first, assessed up to study completion (maximum of 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wei, MBBS, PhD, Principal Investigator — The Alfred
Locations (5):
- Australia (2):
  - The Alfred Hospital, Melbourne
  - Royal Melbourne Hospital, Parkville
- France (3):
  - Institut Paoli Calmettes, Marseille
  - Hôpital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: Yes
Researchers can ask for a study protocol, patient-level and/or study-level clinical trial data including clinical study reports (CSRs).
  They can ask all interventional clinical studies:
  * submitted for new medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * Where Servier or an affiliate are the Marketing Authorization Holders (MAH). The date of the first Marketing Authorization of the new medicine (or the new indication) in one of the EEA Member States will be considered within this scope.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: http://clinicaltrials.servier.com

REFERENCES:
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: study-level clinical trial data — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/